CLINICAL TRIAL: NCT00852943
Title: Screening Protocol for Genetic Diseases of Allergic Inflammation
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090086; 09-I-0086
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-08-29

CONDITIONS: Eosinophilic Disease; Immune Deficiency; HaTS; Urticaria Anaphylaxis; Elevated IgE Level
Keywords: IMMUNODEFICIENCY DISEASES; GENETIC DISEASE; Inherited Allergic Disease; Allergy; Autoimmune Diseases; Natural History
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Genetic Diseases, Inborn; Hypersensitivity; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Subjects, ages birth to 99 years old, known to have or suspected of having an inherited disorder of allergic inflammation or mast cell homeostasis or activation, will be eligible for enrollment.

SUMMARY:
Background:

* Mast cells are responsible for most symptoms of allergic reactions. In some allergic diseases, it is unusually easy to cause mast cells to release their contents and cause allergic reactions. In other cases, mast cells grow abnormally and, in rare cases, can result in tumors. Mast cells also control other parts of the immune system.
* Understanding why mast cells behave abnormally in allergic diseases is important to finding better ways for diagnosing and treating these potentially life-threatening disorders.

Objectives:

* To screen mast cells at the genetic and functional levels to characterize abnormalities, identify mutations, detect carrier states, and/or develop therapies for such disorders.
* To create a library of information about inherited diseases of mast cell homeostasis and activation, including piebaldism (problems with skin and hair pigmentation), anaphylaxis (severe allergic reaction), allergies, asthma, atopic dermatitis (eczema), allergic rhinitis ( hay fever ), food allergies, urticaria/angioedema (hives/swelling), immunodeficiency diseases, and autoimmune diseases.

Eligibility:

* Patients between the ages of 1 and 80 years who have been referred by a physician and are known to have or be suspected of having an inherited disorder of mast cells, in particular patients (and their relatives) with piebaldism, allergies, or anaphylaxis that is not caused by allergies.

Design:

* Study population will consist of up to 1000 participants in a 5-year period. One third of the study population will consist of patients; the other two thirds will consist of biological relatives.
* Evaluation is limited to testing on blood specimens; no treatment will be provided.
* Clinical and research laboratory evaluations of patients will include the following:
* Clinical evaluation and previous laboratory tests as documented in outside medical records by health care providers. A standard questionnaire will also be administered at the time of subject enrollment.
* Blood collection for clinical laboratory testing, tailored to each subject s clinical evaluation where appropriate (5 ml).
* Blood collection for research laboratory testing, tailored to each subject s clinical evaluation including genetic screening and assessment of mast cell growth and functioning and storage of additional frozen blood specimens for future studies (up to an additional 30 ml).
* Evaluations of blood relatives will include the following:
* Clinical evaluation as documented from outside medical records by health care providers and administration of a standard questionnaire.
* Blood collection where indicated for diagnostic or research purposes.
* After 12 consecutive months on the study, results from initial evaluation will be reviewed. Subjects with findings deemed to be of continued interest will be contacted and invited to remain as active participants to this protocol for another year, provided that they renew their consent to participate.

DETAILED DESCRIPTION:
This protocol is designed to screen subjects (and some family members) with suspected or identified genetic diseases of allergic inflammation or mast cell homeostasis and activation. Patients determined by clinical history and initial outside evaluation by their referring physician to be of interest will be consented and enrolled into this study. Blood specimens, stored blood products and derivatives, saliva, hair, fingernail clippings, cord blood, umbilical cord, and/or buccal swabs from such patients and/or their family members will be obtained for research studies related to understanding the genetic and biochemical bases of these diseases. Outside medical records may be obtained for chart review to correlate clinical history to research laboratory testing results. Results will be relayed to the referring physicians and, where applicable, patients will be referred to other appropriate NIH protocols for additional clinical evaluation and treatment. The study will enroll up to 1000 subjects and family members.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects, ages birth to 99 years old, known to have or suspected of having an inherited or acquired genetic disorder resulting in severe allergic inflammation and/or reactivity associated with alterations in mast cell and/or eosinophil homeostasis or activation, will be eligible for enrollment. Because of the intensive time and labor required for research laboratory testing, subjects will be enrolled only if in the opinion of the investigator (based on discussions with the patient s private physician) there is a high index of suspicion of a genetic basis for the observed allergic manifestation(s).
* Blood relatives of enrolled subjects will be eligible for enrollment.
* There will be no discrimination as to age, gender, race, or disability.
* Subjects must have a health care provider outside of the NIH.
* Subjects must agree to have their blood stored for future studies of the immune system and/or other medical conditions.

EXCLUSION CRITERIA:

- Ongoing systemic immune modulation with agents such as biologics that target mast cells and eosinophils, immune modulating or cytotoxic chemotherapy, and/or malignancy may be grounds for possible exclusion if, in the opinion of the investigator, the presence of such a disease process would interfere with evaluation.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Disorders of allergic inflammation and mast cell homeostasis and activation.
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2010-11-02 (Actual)

PRIMARY OUTCOMES:
Association of single gene mutations which are deemed causal with specific syndromic presentations of allergic disease, including atopic dermatitis, asthma, food allergy, eosinophilic disease, urticaria anaphylaxis, angioedema, IgE levels and ch... | end of study or until a gene is found
  Association of single gene mutations which are deemed causal with specific syndromic presentations of allergic disease, including atopic dermatitis, asthma, food allergy, eosinophilic disease, urticaria anaphylaxis, angioedema, IgE levels and changes to allergy-related effector cells.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela A Guerrerio, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-I-0086.html